CLINICAL TRIAL: NCT07189455
Title: A Multicenter, Randomized, Controlled, Open-Label Phase III Study Evaluating the Efficacy and Safety of ZG006 for Injection Compared With Investigator-Selected Chemotherapy in Participants With Relapsed Small Cell Lung Cancer
Brief Title: Study Comparing ZG006 With Investigator-Selected Chemotherapy in Participants With Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-006
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZG006 (Experimental): ZG006 10 mg Q2W
  Interventions: Drug: ZG006
- Investigator-Selected Chemotherapy (Active Comparator): Investigator-selected chemotherapy, such as topotecan.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.
  Arms: ZG006
Drug: Topotecan — Topotecan will be administered per local standard of care
  Arms: Investigator-Selected Chemotherapy

SUMMARY:
The main objective is to compare ZG006 with Investigator-Selected Chemotherapy on prolonging overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years of age;
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months;
* Histologically or cytologically confirmed Small Cell Lung Cancer.

Exclusion Criteria:

* Participants were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3 years

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 3 years
Serum Concentrations of ZG006 | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China